CLINICAL TRIAL: NCT02545465
Title: Retrospective Chart Review of Patients With PAH or Inoperable/Persistent/Recurrent CTEPH Who Transition Their PH Treatment to Adempas
Brief Title: A Study to Understand the Treatment Patterns in Patients With Pulmonary Arterial Hypertension or Chronic Thromboembolic Pulmonary Hypertension During a Switch of Treatment to Adempas in Real-life Clinical Practice
Acronym: CAPTURE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17983; AD1501 (Other: Company Internal)
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension; Inoperable Chronic Thromboembolic Pulmonary Hypertension; Persistent Chronic Thromboembolic Pulmonary Hypertension; Recurrent Chronic Thromboembolic Pulmonary Hypertension; Switch of therapy; Titration phase; Retrospective chart review
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BAY63-2521: Patients who have been switched from a Pulmonary Hypertension treatment to Adempas
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — As per the treating physicians discretion

SUMMARY:
The aim of this study is to understand the treatment patterns in patients with Pulmonary Arterial Hypertension (PAH) or Chronic Thromboembolic Pulmonary Hypertension (CTEPH) during a switch of treatment to Adempas in real-life clinical practice.

In addition, this study will describe patient demographics and reason for switching

ELIGIBILITY:
Inclusion Criteria:

- Female and male adult patients diagnosed with PAH or inoperable/recurrent/persistent CTEPH who have been switched from a PH treatment (i.e. Endothelin Receptor Antagonist(ERAs), Phosphodiesterase-5 inhibitor(PDE5i) or Prostacyclin Analog (PCA) to Adempas

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice
* Patients who have not switched their therapy from an Endothelin Receptor Antagonist (ERA) or Prostacyclin Analog (PCA) but received Adempas purely as an add-on therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Source population of the study are patients with Pulmonary arterial hypertension(PAH) and Chronic thromboembolic pulmonary hypertension (CTEPH). Patients with this rare condition are mostly diagnosed and managed at specialist centers. This includes initiation or any change of Pulmonary Hypertension (PH) therapy. The participation of these specialized centers in the study is going to ensure the representativeness of the study population. In order to reduce selection bias physicians will be asked to include all eligible patients.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Starting Dose | Up to a total of 8 weeks of titration period
Dose Increments | Up to a total of 8 weeks of titration period
Final Dose | Up to a total of 8 weeks of titration period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Many Locations, Belgium
- Many Locations, Canada
- Many Locations, Colombia
- Many Locations, Germany
- Many Locations, Japan
- Many Locations, Sweden
- Many Locations, Turkey (Türkiye)